CLINICAL TRIAL: NCT01510405
Title: Phosphoproteomic Patterns as a Novel Biomarker for Aurora and Polo-like Kinase Inhibitors in Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Konstantin Dragnev, Staff Physician, Hematology-Oncology, Dartmouth-Hitchcock Medical Center
Other Study IDs: D1026
Record Dates: First submitted 2012-01-06; First posted 2012-01-16 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Subjects undergoing or who have undergone thoracic surgery for presumed lung cancer.; The following procedures are allowed: Wedge resection, lobectomy, bilobectomy, segmentectomy and pneumonectomy thoracic surgical operations are permitted.
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Tissue Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 40 Participants: Participants undergoing or who have undergone thoracic surgery for presumed lung cancer with a wedge resection, lobectomy, bilobectomy, segmentectomy and/ or pneumonectomy thoracic surgical operation.
  Interventions: Other: Tissue Collection

INTERVENTIONS:
Other: Tissue Collection — Tissue sample collection
  Other Names: Frozen tissue specimens will be stored at -80

SUMMARY:
The investigators have characterized in preclinical Non-Small Cell Lung Cancer (NSCLC) models the proteomic expression profile associated with exposure to Aurora and Polo-like kinase inhibitors. The identification of proteomic expression patterns in patients with NSCLC would be an important step in defining the possible role of these agents as potential targeted therapies for this clinically important disease. This study proposes to evaluate resected non-small cell lung cancer specimens for these proteomic expression profiles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing or who have undergone thoracic surgery for presumed lung cancer
* Wedge resection, lobectomy, bilobectomy, segmentectomy and pneumonectomy thoracic surgical operations are permitted.
* Age ≥ 18 years.
* Subject meets criteria for thoracic surgery as determined by the thoracic surgeon.
* Able to provide written informed consent.

Exclusion Criteria:

* Subjects undergoing or who have undergone thoracic surgery for metastatic disease from other primary sources such as colorectal cancer, sarcoma, melanoma, breast cancer, bladder cancer, prostate cancer, esophageal cancer, pancreatic cancer, or gastric cancer will be excluded.
* Subjects who have received prior preoperative lung cancer anticancer therapy will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have presumed lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2010-07; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Correlation between the Phosphoproteomic expression pattern of specific substrates of Aurora Kinase A and/or Polo-like kinase 1 (PLK1) | 2 years
  Correlation of phosphoproteomic expression patterns of specific substrates of Aurora kinase A and/or Polo-like kinase 1 and disease-free survival in surgically resected NSCLC. (Disease-free survival is defined as the time from surgical resection until the first documentation of disease recurrence or death.)

SECONDARY OUTCOMES:
Phosphoproteomic Expression Profiles and Correlated Global Phosphoproteomics Expression patterns | 2 years
  To establish and validate a technology for quantitatively determining global phosphoproteomic expression profiles in surgically resected NSCLC specimens and To correlate global phosphoproteomics expression patterns with time to disease recurrence, lung cancer-specific survival and overall survival.
Time to Disease Recurrence | 2 years
  Time to disease recurrence: Correlation of phosphoroteomic expression patterns of specific substrates of Aurora Kinase A and/or Polo-like kinase 1 and time to disease recurrence defined as the time from surgical resection until the first documented evidence of disease recurrence
Lung Cancer Specific Survival | 2 years
  Correlation of phosphoproteomic expression patterns of specific substrates of Aurora kinase A and/or Polo-kinase 1 and lung cancer specific survival defined as the time from surgical resection until death from lung cancer. For subjects who have died from other causes than lung cancer, time to death will be censored at the time of death from causes other than lung cancer.
Overall Survival | 2 Years
  Correlation of phosphproteomic expression patters of specific substrates of Aurora kinase A and/or Polo-like kinase 1 and overall survival defined as the time from surgical resection until death due to any cause. For subjects who do not yet die, time to death will be censored at the time of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: James R Rigas, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States